CLINICAL TRIAL: NCT07266233
Title: Evaluation of the Antibacterial Activity and Postoperative Pain Outcomes of Photodynamic Therapy Using Toluidine Blue
Brief Title: Toluidine Blue-Based Photodynamic Therapy for Antibacterial Activity and Postoperative Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, AZİZ ŞAHİN ERDOĞAN, Assistant Professor, Department of Endodontics, Faculty of Dentistry, Atatürk University, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AU-DHF-ASE-01
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Root Canal Infection
MeSH Terms: interventions — Tolonium Chloride; Photochemotherapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups (experimental and control) and will receive the allocated intervention only. Each participant will remain in the assigned group for the duration of the study.
Who Masked: Participant
Masking Description: A single-blind design was implemented. Participants were unaware of their assigned intervention, and outcome assessors performing the microbiological analysis were masked to group allocation. A sham light application was used in the control group to preserve blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham PDT) (Placebo Comparator): Participants in this arm will receive the standard root canal irrigation protocol using 2.5% sodium hypochlorite and 17% EDTA. A sham photodynamic procedure will be performed by positioning the LED device near the tooth without light activation to simulate photodynamic therapy conditions. No Toluidine Blue O will be applied, and no active light irradiation will be performed
  Interventions: Procedure: Sham Photodynamic Therapy
- Experimental Group (PDT) (Experimental): Participants in this arm will receive the standard root canal irrigation protocol followed by adjunctive photodynamic therapy. A 0.1 mg/mL Toluidine Blue O solution will be delivered into the canal and activated with a 630-nm LED light using an optical fiber for 60 seconds. This procedure will be performed after instrumentation and prior to final assessment sampling.
  Interventions: Drug: Toluidine Blue O (0.1 mg/mL); Device: 630-nm LED Light Device; Procedure: Photodynamic Therapy (PDT)

INTERVENTIONS:
Drug: Toluidine Blue O (0.1 mg/mL) — A 0.1 mg/mL toluidine blue O solution used as the photosensitizer for photodynamic therapy. The solution is placed into the root canal prior to 630-nm LED irradiation for activation.
  Arms: Experimental Group (PDT)
Device: 630-nm LED Light Device — A light-emitting diode device delivering 630-nm wavelength used to activate toluidine blue O during photodynamic therapy. The device is positioned near the tooth for 60 seconds.
  Arms: Experimental Group (PDT)
Procedure: Photodynamic Therapy (PDT) — Application of 0.1 mg/mL toluidine blue O into the root canal, followed by activation with a 630-nm LED light source for 60 seconds as part of the experimental disinfection protocol.
  Arms: Experimental Group (PDT)
Procedure: Sham Photodynamic Therapy — Placebo photodynamic procedure in which the LED device is positioned similarly but activated without delivering light energy; no toluidine blue O is applied.
  Arms: Control Group (Sham PDT)

SUMMARY:
This clinical study aims to evaluate the antimicrobial effectiveness and postoperative pain outcomes of photodynamic therapy using Toluidine Blue O as an adjunct to conventional root canal treatment in patients diagnosed with symptomatic irreversible pulpitis. Photodynamic therapy is a non-invasive light-activated disinfection method, and this study will compare its performance with standard endodontic treatment protocols. The results are expected to provide clinical evidence regarding its potential benefits in reducing intracanal bacterial load and improving postoperative patient comfort.

DETAILED DESCRIPTION:
This randomized clinical study is designed to investigate the antimicrobial effectiveness and postoperative pain outcomes of photodynamic therapy (PDT) using toluidine blue O (TBO) as an adjunct to conventional root canal treatment in single-rooted teeth with necrotic pulps. The rationale for this research is based on the persistent difficulty of achieving complete microbial elimination from the root canal system using standard chemomechanical preparation alone. Toluidine blue O-mediated PDT has been proposed as a minimally invasive disinfection method capable of producing reactive oxygen species after activation with visible light, thereby enhancing microbial reduction beyond that achieved by irrigation protocols.

The study employs a standardized protocol in which intracanal microbiological sampling is conducted at four predefined stages to monitor changes in microbial load throughout treatment. All samples are stored and analyzed using real-time quantitative polymerase chain reaction (qPCR), which allows sensitive detection and quantification of bacterial DNA. This molecular approach offers advantages over culture-based methods by identifying uncultivable or low-abundance bacterial species, providing a more comprehensive evaluation of the antimicrobial effect of PDT.

In the experimental group, photodynamic therapy is performed by introducing a 0.1 mg/mL toluidine blue O solution into the prepared root canal, followed by activation with a 630-nm LED light source. The choice of this wavelength corresponds to the absorption peak of TBO and optimizes energy transfer for singlet oxygen production. A sham procedure is used in the control group to maintain participant masking and ensure methodological consistency. Both groups receive identical chemomechanical preparation and irrigation procedures prior to the assigned intervention.

Pain assessment during the postoperative period is performed using a validated visual analog scale (VAS), providing continuous measurement of patient-reported discomfort during the first week after treatment. The integration of molecular microbiology with clinical pain evaluation allows a combined assessment of both biological and patient-centered outcomes. This study is expected to contribute new in-vivo evidence on the potential benefits of toluidine blue O-based PDT as an adjunctive disinfection method in endodontic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 65 years
2. Presence of asymptomatic apical periodontitis with necrotic pulp in single-rooted maxillary or mandibular incisors, canines, or premolars
3. Periapical Index (PAI) score ≥ 2
4. Patients classified as ASA I (American Society of Anesthesiologists Physical Status Classification)
5. Preoperative pain score < 50 on the Visual Analog Scale (VAS)

Exclusion Criteria:

1. Multi-rooted teeth
2. Patients classified as ASA II or higher
3. Pregnant women or those with suspected pregnancy
4. Root canal curvature greater than 25° according to the Schilder method
5. Patients diagnosed with generalized periodontitis
6. Periodontal pocket depth > 3 mm in the related tooth
7. Use of analgesic medication within the past 72 hours
8. Use of antibiotic therapy within the past month
9. Presence of swelling and positive response to palpation/percussion tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in intracanal bacterial load measured by quantitative PCR (qPCR) | Baseline (Day 1) to Immediately After Intervention (Day 1)
  Intracanal bacterial load will be quantified using real-time quantitative polymerase chain reaction (qPCR). Samples will be collected at four predefined sampling points (S0-S3) using sterile #30 paper points inserted into the canal for 30 seconds.
  S0 (Baseline): After isolation and disinfection, before instrumentation
  S1: After access cavity preparation and working length determination
  S2: After root canal instrumentation
  S3 (Post-Intervention): After final irrigation protocol and photodynamic therapy (or sham procedure)
  Changes in bacterial DNA concentration (copy number/µL) from S0 to S3 will be compared between groups.

SECONDARY OUTCOMES:
Postoperative pain levels measured using the Visual Analog Scale (VAS, 0-100) | 6 hours, 12 hours, 24 hours, Day 3, Day 5, and Day 7 after treatment.
  Postoperative pain intensity will be measured using the Visual Analog Scale (VAS), a 100-mm line ranging from 0 to 100, where 0 represents "no pain" and 100 represents "worst imaginable pain." Higher scores indicate worse pain. Participants will record their pain levels at each scheduled assessment time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Faculty of Dentistry, Department of Endodontics, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Er Karaoglu G, Ugur Ydin Z, Erdonmez D, Gol C, Durmus M. Efficacy of antimicrobial photodynamic therapy administered using methylene blue, toluidine blue and tetra 2-mercaptopyridine substituted zinc phthalocyanine in root canals contaminated with Enterococcusaecalis. Photodiagnosis Photodyn Ther. 2020 Dec;32:102038. doi: 10.1016/j.pdpdt.2020.102038. Epub 2020 Oct 1. PMID 33010484
- [Background] Mozayeni MA, Vatandoost F, Asnaashari M, Shokri M, Azari-Marhabi S, Asnaashari N. Comparing the Efficacy of Toluidine Blue, Methylene Blue and Curcumin in Photodynamic Therapy Against Enterococcus faecalis. J Lasers Med Sci. 2020 Fall;11(Suppl 1):S49-S54. doi: 10.34172/jlms.2020.S8. Epub 2020 Dec 30. PMID 33995969